CLINICAL TRIAL: NCT00056329
Title: Multicenter Vitamin E Trial in Aging Persons With Down Syndrome
Brief Title: Vitamin E in Aging Persons With Down Syndrome
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: New York State Institute for Basic Research (Other Government)
Collaborators: National Institute on Aging (NIA) (NIH); Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH); National Center for Complementary and Integrative Health (NCCIH) (NIH)
Responsible Party: Principal Investigator, Arthur Dalton, Deputy Director, New York State Institute for Basic Research
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: IA0039; R01AG016381 (NIH); NIA Grant AG16381
Record Dates: First submitted 2003-03-10; First posted 2003-03-12 (Estimated); Last update posted 2012-05-04 (Estimated); Status verified 2012-05

CONDITIONS: Down Syndrome; Alzheimer Disease
Keywords: Aging Persons; Down Syndrome; Vitamin E; Alzheimer disease
MeSH Terms: conditions — Down Syndrome; Alzheimer Disease | interventions — Vitamin E; Tocopherols; Geritol

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Experimental): vitamin E plus multivitamin
  Interventions: Drug: Vitamin E; Drug: multivitamin
- 2 (Placebo Comparator): placebo with multivitamin
  Interventions: Drug: multivitamin; Drug: Placebo

INTERVENTIONS:
Drug: Vitamin E — 1,000 international units twice daily for three years
  Other Names: tocopherol
  Arms: 1
Drug: multivitamin — once daily for three years
Drug: Placebo — Placebo twice daily for three years
  Arms: 2

SUMMARY:
The goal of this study is to determine the safety and efficacy of the administration of vitamin E, which has been shown to delay the progression of Alzheimer's disease, in slowing the rate of cognitive/functional decline in older persons with Down syndrome.

DETAILED DESCRIPTION:
The growing success of therapeutic interventions (including the antioxidant Vitamin E) for Alzheimer's disease in the general population requires a solution to the methodological problems so that therapeutic trials can be conducted in the aging population with Down syndrome which will ultimately improve their quality of life as well as that of their families and caregivers. The experience gained in this trial will be useful to the design of appropriate cognitive measures of Alzheimer's disease in persons with Down syndrome in subsequent trials.

The goal of this international three-year study is to determine whether the administration of vitamin E, which has been shown to delay the progression of Alzheimer's disease, will slow the rate of cognitive/functional decline in persons age 50 or older with Down syndrome. Persons with Down syndrome functioning at all levels of intellectual disability will be eligible. Men and women of approximately equal numbers and people from minorities and ethnic groups other than Caucasian will be included. A total of 350 individuals with Down syndrome, 50 years of age and older, have been recruited at approximately 21 trial sites. The study is a randomized, double-blind, placebo-controlled, parallel group design with stratification by geographic site and presence of Alzheimer disease according to DSM-IV (American Psychiatric Association) criteria for diagnosing this disease.

Apolipoprotein E (Apo E) genotype will be determined at the screening visit to allow secondary analyses of the impact of Apo E genotype (that may influence Alzheimer's disease risk) on outcome measures and the response to treatment. DNA specimens will also be stored for possible future genetic analyses, with trial sites allowing for non-participation in this procedure. Visits will occur at baseline and then at 6 monthly intervals, with each visit including interval medical history, current and interval medications, side effects checklist, adverse events, pill count, institutionalization status, cognitive, functional, and behavioral measures, and DSM-IV diagnostic assessment for Alzheimer's disease.

ELIGIBILITY:
Inclusion Criteria:

* Presence of clinically determined Down syndrome (karyotypes optional).
* Medically stable.
* Medications stable over 3 months.
* Appropriately signed and witnessed consent form.
* Involvement/cooperation of informant/caregiver.

Exclusion Criteria:

* Medical/neurological condition (other than Alzheimer's disease) associated with dementia.
* Brief Praxis Test score <20.
* Modified Hachinski score >4.
* Major depression within 3 months.
* History of any disorder of blood coagulation (inherited or acquired).
* Current use of anti-coagulants.
* Use of experimental medications within 3 months.
* Regular use of vitamin E greater than 50 units per day during the previous 6 months.

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 350 (Actual)
Dates: Start 2002-04; Primary Completion 2012-05 (Estimated); Study Completion 2012-05 (Estimated)

PRIMARY OUTCOMES:
Brief Praxis Test, measuring cognitive functions expressed as performances of simple, short, sequences of voluntary movements | Screening, Baseline, every 6 months for 36 months

SECONDARY OUTCOMES:
Fuld Object Memory Test (Modified), New Dot Test, Orientation Test, Vocabulary Test, Behavior & Function Down Syndrome Rating Scale, Clinical Global Impression of Change (CGI-C) | Screening, Baseline, and every 6 months for 36 months

CONTACTS AND LOCATIONS:
Overall Officials: Arthur J Dalton, PhD, Principal Investigator — New York State Institute for Basic Research in Developmental Disabilities; Paul S Aisen, MD, Study Director — Georgetown University; Mary C Sano, PhD, Study Director — Icahn School of Medicine at Mount Sinai
Locations (22):
- United States (14):
  - University of Connecticut Health Center, Farmington, Connecticut
  - Roskamp Institute Memory Clinic, Tampa, Florida
  - Institute for the Study of Disadvantage and Disability, Atlanta, Georgia
  - May South, Inc., Atlanta, Georgia
  - University of Illinois at Chicago, Chicago, Illinois
  - Southern Illinois University School of Medicine, Springfield, Illinois
  - Third Age, Inc., Lexington, Kentucky
  - McLean Hospital, Belmont, Massachusetts
  - Clinical Research Center of New Jersey, Voorhees Township, New Jersey
  - University at Albany, SUNY, Albany, New York
  - Nathan Kline Institute, Orangeburg, New York
  - George Jervis Clinic, Staten Island, New York
  - Westchester Institute for Human Development, Valhalla, New York
  - University Memory and Aging Center, Case Western Reserve University, Cleveland, Ohio
- Centre for Developmental Disabilities Studies, Ryde, New South Wales, Australia
- Canada (3):
  - Down Syndrome Research Foundation, Port Coquitlam, British Columbia
  - Surrey Place Centre, Toronto, Ontario
  - Saskatoon City Hospital, Saskatoon, Saskatchewan
- United Kingdom (4):
  - University of Cambridge, Cambridge, England
  - Greenfields Monyhull Hospital, Kings Norton, Birmingham, England
  - Kings College: London, London, England
  - Mercer Institute for Research on Ageing, St. James Hospital, Dublin, Ireland

REFERENCES:
- [Background] Sano M, Ernesto C, Thomas RG, Klauber MR, Schafer K, Grundman M, Woodbury P, Growdon J, Cotman CW, Pfeiffer E, Schneider LS, Thal LJ. A controlled trial of selegiline, alpha-tocopherol, or both as treatment for Alzheimer's disease. The Alzheimer's Disease Cooperative Study. N Engl J Med. 1997 Apr 24;336(17):1216-22. doi: 10.1056/NEJM199704243361704. PMID 9110909
- [Background] Aisen PS, Davis KL. The search for disease-modifying treatment for Alzheimer's disease. Neurology. 1997 May;48(5 Suppl 6):S35-41. doi: 10.1212/wnl.48.5_suppl_6.35s. PMID 9153159
- [Background] Aylward EH, Burt DB, Thorpe LU, Lai F, Dalton A. Diagnosis of dementia in individuals with intellectual disability. J Intellect Disabil Res. 1997 Apr;41 ( Pt 2):152-64. doi: 10.1111/j.1365-2788.1997.tb00692.x. PMID 9161927
- [Background] Dalton, AJ, Mehta, PD, Fedor, BL, Patti, PJ: Cognitive changes in memory precede those in praxis in aging persons with Down syndrome. Journal of Intellectual and Developmental Disability 24(2):169-187,1999.
- [Result] Sano M, Aisen PS, Dalton AJ, Andrews HF, Tsai W-Y, and the International Down Syndrome Alzheimer Disease Consortium. Assessment of aging individuals with Down syndrome in clinical trials: results of baseline measures. Journal of Policy and Practice in Intellectual Disabilities. 2005 2(2):126-138.